CLINICAL TRIAL: NCT06585085
Title: Care Pathway Organization in Order to Increase Physical Activity Levels and Limit Sedentary Behavior During Pregnancy: a Randomized Controlled Trial
Brief Title: Physical Activity and Sedentary Behavior During Pregnancy
Acronym: PREGMOUV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Réseau de Santé en Périnatalité d'Auvergne (Unknown); ASM Omnisports - Pôle Sport-Santé (Unknown); Office Municipal du Sport - Espace Sport Santé (Unknown); Observatoire national de l'activité physique et de la sédentarité (Unknown); Ville de Clermont-Ferrand (Unknown); Ministère de la Santé et de la Prévention (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: RBHP 2024 BARASINSKI; 2024-A00459-38 (Other: ANSM)
Record Dates: First submitted 2024-08-26; First posted 2024-09-05 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Pregnant Woman
Keywords: physical activity; sedentary behaviour; care pathway
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- A - Free PA practice (No Intervention): The women in group A (control group) will receive the usual care provided for any pregnancy, i.e. personalised information on physical activity and sedentary behaviour, with the provision of information booklets. They will be free to exercise during their pregnancy
- B (Experimental): In-person supervised PA sessions
  Interventions: Behavioral: In person PA sessions
- C (Experimental): Interactive videoconference PA sessions
  Interventions: Behavioral: Interactive videoconference PA sessions
- D (Experimental): In person and by videoconference (mixed format) PA sessions
  Interventions: Behavioral: In person and by videoconference (mixed format) PA sessions.

INTERVENTIONS:
Behavioral: In person PA sessions — Group B women will have access to a weekly program of 3 face-to-face PA sessions. The face-to-face sessions will be offered at one or more locations in the Clermont-Ferrand area, depending on the number of groups taking part. They will also be offered at one or more times depending on the number of groups. Locations and times will be specified on the online booking software. Women can only register for 3 sessions per week.
  Arms: B
Behavioral: Interactive videoconference PA sessions — Women in Group C will have access to a weekly program of 3 PA sessions via interactive videoconferencing. These sessions will have the same format as the face-to-face sessions with visualization of the APA professional, visualization of the participants (who can also choose to be masked). The PA professional will also see the participants, so he or she can correct positions and give individualized advice at any time. Schedules will be specified on the online booking software with the videoconference link. Women can only register for 3 sessions per week.
  Arms: C
Behavioral: In person and by videoconference (mixed format) PA sessions. — Women in Group D will have access to a weekly program of 3 mixed-format PA sessions, with 2 interactive distance learning sessions and 1 in-person session. The in-person sessions will be offered at one or more locations in the Clermont-Ferrand area, depending on the number of groups taking part. Locations and times will be specified on the online booking software. Women can only register for 1 face-to-face session per week. The other 2 sessions will be offered via interactive videoconferencing. These sessions will have the same format as the in-person sessions, with visualization of the APA professional, visualization of the participants. The APA professional will also see the participants, so he or she can correct positions and give individualized advice at any time. Schedules will be specified on the online booking software with the videoconference link. Women can only register for 2 videoconference's sessions per week.
  Arms: D

SUMMARY:
Our main objective is to evaluate the intervention that best enables women's adherence to physical activity (PA).

Our hypothesis is that identifying types of interventions suitable for pregnant women (in-person PA sessions, videoconferences or mixed format) could help improve their PA level and simultaneously reduce their sedentary behavior (SB).

DETAILED DESCRIPTION:
PA has beneficial effects on physical, psychological, and social health, and its regular practice helps to prevent numerous chronic diseases. During pregnancy, PA also has many benefits for women's physical condition, weight gain, gestational hypertension, lower back and pelvic pain, and postpartum depressive symptoms and may also reduce fetal macrosomia and positively affect neurogenesis, language development, memory, and other learning-associated cognitive functions. (CNSF 2021). PA is thus recommended to all pregnant women for 150 to 180 minutes a week, adapted to their health status, physical condition, and course of pregnancy. It is also recommended that women limit their Sedentary Behaviour (SB) (to ≤7 waking h/day) during pregnancy.

No French study has assessed the impact of a PA program during pregnancy, and no published study has proposed videoconference PA sessions during pregnancy. Pregnant women's adherence to PA is a limiting factor found in many interventional studies. Possible changes in maternal behavior in practicing PA and reducing SB during pregnancy could also favorably affect the health of mother and child and thus subsequent PA. Given PA's many benefits and SB's harmful effects during pregnancy, assessing programs that enable pregnant women to both increase PA levels and reduce SB seems pertinent and valuable.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women of more of 18 years and who are being monitored for pregnancy in the Clermont-Ferrand metropolitan area,
* Planned to give birth in a maternity unit localized in Clermont-Ferrand metropolitan area (CHU Estaing or Clinique de la Chataigneraie),
* Agreeing to be randomized, to follow the physical activity program offered in the Clermont-Ferrand metropolitan area, and to follow up as part of the study,
* Able to give informed consent to participate in the research,
* Affiliated to a social security scheme
* And between 14+0d and 21+6d weeks of gestation.

Non inclusion Criteria:

* Women under guardianship, curators, deprived of liberty or under court protection,
* With a history of recurrent miscarriage,
* Presenting a multiple pregnancy,
* Hemoglobinemia <9g/dL or symptomatic anemia,
* Presenting eating disorders or a BMI ≤ 18.5 or a BMI ≥ 40,
* With orthopedic limitations,
* Presenting cardiovascular or pulmonary disease,
* Uncontrolled thyroid disease,
* Presenting a high level of smoking,
* With significant health problems,
* Premature rupture of membranes,
* Premature labor during this pregnancy or a history of at least 2 premature births,
* Persistent vaginal bleeding,
* Cervical incompetence,
* Evidence of intrauterine growth restriction,
* Uncontrolled epilepsy,
* Diabetes (previous or gestational, diagnosed in the 1st trimester) or chronic hypertension,
* Or having a planned home birth.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Study focused on pregnant women
Enrollment: 630 (Estimated)
Dates: Start 2024-09-10 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Women's adherence to PA at the end of the second trimester | between 24 and 30 weeks of gestation
  measurement of the PA level, measured by accelerometer, expressed in MET.minutes/week by wearing a tri-axial accelerometer on the hip

SECONDARY OUTCOMES:
women's adherence in terms of reduction of Sedentary Behaviors at the end of the 2nd trimester | between 24 and 30 weeks of gestation
  measurement of sedentary time (defined as a state of wakefulness characterized by an energy expenditure less than or equal to 1.5 METs) between getting up and going to bed using a tri-axial hip accelerometer
Women's participation at PA sessions | After 39 weeks of gestation, end of planned participation in sessions
  For women in groups B, C and D, rate of sessions completed on the number of eligible sessions according to their randomization group and the socio-demographic criteria
Pregnancy and Postpartum Evolution of PA Time | at 4 distinct times: between 24+0d and 30+0d weeks of gestation, between 32+0d and 37+6d weeks of gestation, between 6 and 10 weeks postpartum and between 20 and 24 weeks postpartum
  PA time measured with a tri-axial accelerometer at the hip
Evolution in sedentary behavior during pregnancy and postpartum | at 4 distinct times: between 24 and 30 weeks of gestation, between 32+0day and 37+6day weeks of gestation, between 6 and 10 weeks postpartum and between 20 and 24 weeks postpartum
  sedentary time (defined as wakefulness characterized by an energy expenditure less than or equal to 1.5 METs) between getting up and going to bed will be compared according to each intervention modality. Sedentary behavior will be measured by wearing a tri-axial accelerometer on the hip
Women's perception of the determinants of their level of physical activity and sedentary behaviour | during the 31 days after at the inclusion in the study and between 35 and 39 weeks of gestation
  Qualitative study by means of semi-structured telephone interviews with a minimum of 100 women, i.e. a minimum of 25 women per group, a number to be adapted according to the data saturation that will be obtained
Impact of physical activity on maternal antenatal morbidity | At delivery
  occurrence of maternal pathology during pregnancy (gestational arterial hypertension [PAS ≥ 140 mm Hg and a PAD ≥ 90 mm Hg occurring after 20 weeks of gestation] and/or, pre-eclampsia [hypertension with albuminuria > 0.3g/L per 24 hours] and/or gestational diabetes diagnosed by orally induced hyperglycaemia after 23 SA)
Impact of sedentary behaviour on maternal antenatal morbidity | At delivery
  occurrence of maternal pathology during pregnancy (gestational arterial hypertension [PAS ≥ 140 mm Hg and a PAD ≥ 90 mm Hg occurring after 20 weeks of gestation] and/or, pre-eclampsia [hypertension with albuminuria > 0.3g/L per 24 hours] and/or gestational diabetes diagnosed by orally induced hyperglycaemia after 23 SA)
Impact of physical activity on perpartum maternal morbidity | 24 hours after delivery
  A composite criterion: "occurrence of 3rd or 4th degree perineal lesions and/or occurrence of immediate postpartum haemorrhage (blood loss > 500mL in the 24 hours after delivery)"
Impact of sedentary behaviour on perpartum maternal morbidity | 24 hours after delivery
  A composite criterion: "occurrence of 3rd or 4th degree perineal lesions and/or occurrence of immediate postpartum haemorrhage (blood loss > 500mL in the 24 hours after delivery)"
Impact of physical activity on postpartum maternal morbidity | 6 months postpartum
  : presence of a depressive state assessed by the Edinburgh Depression Scale (EPDS) (with a discriminant threshold of the EPDS ≥ 11)
Impact of sedentary behaviour on postpartum maternal morbidity | 6 months postpartum
  : presence of a depressive state assessed by the Edinburgh Depression Scale (EPDS) (with a discriminant threshold of the EPDS ≥ 11)
Impact of physical activity on the experience of childbirth | 4 weeks postpartum
  Evaluation using the Questionnaire for Assessing the Childbirth Experience (QACE)
Impact of sedentary behaviour on the experience of childbirth | 4 weeks postpartum
  Evaluation using the Questionnaire for Assessing the Childbirth Experience (QACE)
Impact of physical activity on the quality of life of pregnant women at the end of the 2nd trimester of pregnancy | between 24 and 30 weeks of gestation
  Score obtained in the WHOQOL-Bref questionnaire
Impact of sedentary behaviour on the quality of life of pregnant women at the end of the 2nd trimester of pregnancy | between 24 and 30 weeks of gestation
  Score obtained in the WHOQOL-Bref questionnaire
Impact of physical activity on the quality of life of pregnant women at the end of the 3rd trimester of pregnancy | between 32 and 37 SA+6day weeks of gestation
  Score obtained in the WHOQOL-Bref questionnaire
Impact of sedentary behaviour on the quality of life of pregnant women at the end of the 3rd trimester of pregnancy | between 32 and 37 SA+6day weeks of gestation
  Score obtained in the WHOQOL-Bref questionnaire
Impact of physical activity on the quality of life of pregnant women at 2 months postpartum | between 6 and 10 weeks postpartum
  Score obtained from the WHOQOL-Bref questionnaire
Impact of sedentary behaviour on the quality of life of pregnant women at 2 months postpartum | between 6 and 10 weeks postpartum
  Score obtained from the WHOQOL-Bref questionnaire
Impact of physical activity on the quality of life of pregnant women at 6 months postpartum | between 20 and 24 weeks postpartum
  Score obtained from the WHOQOL-Bref questionnaire
Impact of sedentary behaviour on the quality of life of pregnant women at 6 months postpartum | between 20 and 24 weeks postpartum
  Score obtained from the WHOQOL-Bref questionnaire
Impact of physical activity on the occurrence of urinary incontinence in the 2nd trimester of pregnancy | between 24 and 30 weeks of gestation
  ICIQ-SF questionnaire score - International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form
Impact of sedentary behaviour on the occurrence of urinary incontinence in the 2nd trimester of pregnancy | between 24 and 30 weeks of gestation
  ICIQ-SF questionnaire score - International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form
Impact of physical activity on the occurrence of urinary incontinence in the 3rd trimester of pregnancy | between 32 and 37 SA+6day weeks of gestation
  ICIQ-SF questionnaire score - International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form
Impact of sedentary behaviour on the occurrence of urinary incontinence in the 3rd trimester of pregnancy | between 32 and 37 SA+6day weeks of gestation
  ICIQ-SF questionnaire score - International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form
Impact of physical activity on the occurrence of urinary incontinence at 6 months postpartum | between 20 and 24 weeks postpartum
  Score on the ICIQ-SF questionnaire - International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form
Impact of sedentary behaviour on the occurrence of urinary incontinence at 6 months postpartum | between 20 and 24 weeks postpartum
  Score on the ICIQ-SF questionnaire - International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form
Impact of physical activity on sexual quality of life | between 20 and 24 weeks postpartum
  Score on the FSFI Female Sexual Function Index questionnaire
Impact of sedentary behaviour on sexual quality of life | between 20 and 24 weeks postpartum
  Score on the FSFI Female Sexual Function Index questionnaire
Impact of physical activity on early neonatal morbidity | At delivery
  a composite criterion: "Apgar score <7 at 5 min and/or arterial pH <7.10 and/or transfer and/or intra-hospital transfer to a neonatal unit"
Impact of sedentary behaviour on early neonatal morbidity | At delivery
  a composite criterion: "Apgar score <7 at 5 min and/or arterial pH <7.10 and/or transfer and/or intra-hospital transfer to a neonatal unit"
Impact of physical activity on the newborn's birth weight | At delivery
  occurence of large for gestational age newborns (birth weight greater than the 95th percentile according to gestational age according to Audipog curves)
Impact of sedentary behaviour on the newborn's birth weight | At delivery
  occurence of large for gestational age newborns (birth weight greater than the 95th percentile according to gestational age according to Audipog curves)
Cost-effectiveness analysis from the point of view of health insurance of the proposed intervention methods | Data collected during the pregnancy and until 2 month of post-partum
  Cost-effectiveness incremental study (including modelling of the gains linked to the reduction in C-section)
cost-utility study analysis from the point of view of health insurance of the proposed intervention methods | Data collected during the pregnancy and until 6 month of post-partum
  Cost-utility study (based on the usefulness felt by women) from the point of view of health insurance using the EQ5D-5L (5 Level Euroqol 5 Dimensions) and a mapping analysis of the WHOQOL-Bref

CONTACTS AND LOCATIONS:
Overall Officials: Chloé BARASINSKI, Principal Investigator — CHU de Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France

IPD SHARING:
Plan to Share IPD: No